CLINICAL TRIAL: NCT04169373
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind Program to Evaluate Efficacy and Safety of Upadacitinib in Adult Subjects With Axial Spondyloarthritis Followed by a Remission-Withdrawal Period
Brief Title: A Study to Evaluate Efficacy and Safety of Upadacitinib in Adults With Axial Spondyloarthritis
Acronym: SELECT-AXIS 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-944; 2022-501018-78-00 (Other: EU CT)
Record Dates: First submitted 2019-11-18; First posted 2019-11-19 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Spondyloarthritis
Keywords: Upadacitinib; Axial Spondyloarthritis (axSpA); Spondyloarthritis; Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylarthritis; Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Study 1: Upadacitinib 15 mg (Experimental): Participants receive 15 mg upadacitinib orally once a day for 104 weeks. Participants who flare after 104 weeks will receive open-label upadacitinib once daily from the time of flare for 24 weeks (re-treatment).
  Interventions: Drug: Upadacitinib
- Study 1: Placebo (Placebo Comparator): Participants receive matching placebo for 14 weeks and then switch to receive 15 mg upadacitinib orally once a day for 90 weeks. Participants who flare after 104 weeks will receive open-label upadacitinib once daily from the time of flare for 24 weeks (re-treatment).
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Study 2: Upadacitinib 15 mg (Experimental): Participants receive 15 mg upadacitinib orally once a day for 104 weeks. Participants who flare after 104 weeks will receive open-label upadacitinib once daily from the time of flare for 24 weeks (re-treatment).
  Interventions: Drug: Upadacitinib
- Study 2: Placebo (Placebo Comparator): Participants receive matching placebo for 52 weeks and then switch to receive 15 mg upadacitinib orally once a day for 52 weeks. Participants who flare after 104 weeks will receive open-label upadacitinib once daily from the time of flare for 24 weeks (re-treatment).
  Interventions: Drug: Upadacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib tablet administered orally
  Other Names: ABT-494; RINVOQ
Drug: Placebo — Placebo for upadacitinib tablet administered orally
  Arms: Study 1: Placebo; Study 2: Placebo

SUMMARY:
This protocol includes 2 standalone studies with randomization, data collection, analysis and reporting conducted independently.

The main objectives of this protocol are:

* To evaluate the efficacy of upadacitinib compared with placebo on reduction of signs and symptoms in adults with active axial spondyloarthritis (axSpA) including biologic disease-modifying antirheumatic drug inadequate responders (bDMARD-IR) ankylosing spondylitis (AS) (Study 1) and non-radiographic axial spondyloarthritis (nr-axSpA) (Study 2).
* To assess the safety and tolerability of upadacitinib in adults with active axSpA including bDMARD-IR AS (Study 1) and nr-axSpA (Study 2).
* To evaluate the safety and tolerability of upadacitinib in extended treatment in adult participants with active axSpA including bDMARD-IR AS who have completed the Double-Blind Period (Study 1) and nr-axSpA who have completed the Double-Blind Period (Study 2).
* To evaluate the maintenance of disease control after withdrawal of upadacitinib.

DETAILED DESCRIPTION:
Study 1 (bDMARD-IR AS) is comprised of a 14-week randomized, double-blind, parallel-group, placebo-controlled period (the Double-Blind Period); a 90-week open-label, long-term extension period (the Open-Label Extension Period); and a 30-day Follow-Up Visit (F/U Visit).

Study 2 (nr-axSpA) is comprised of a 52-week randomized, double-blind, parallel-group, placebo-controlled period (the Double-Blind Period); a 52-week open-label, long-term extension period (the Open-Label Extension Period); and a 30-day F/U Visit.

In the Double-Blind Period for both studies, participants are randomized in a 1:1 ratio to receive either upadacitinib or placebo once daily (QD).

Participants in the placebo group switch to upadacitinib 15 mg QD at Week 14 in the Open-Label Extension Period for Study 1 (bDMARD-IR AS) and Week 52 in the Open-Label Extension Period for Study 2 (nr-axSpA).

Participants in remission at Week 104 have the option to enroll in a remission-withdrawal period.

Study M19-944 protocol uses a common screening platform for determining eligibility into Study 1 and Study 2. Each study has its own objectives, hypothesis testing, randomization, data collection, and adequate power for primary and secondary endpoints. Analysis and reporting are conducted separately and independently for each study.

ELIGIBILITY:
Inclusion Criteria:

* Study 1:

  * Must have a clinical diagnosis of ankylosing spondylitis (AS) and meet the modified New York Criteria for AS,
  * Must not have total spinal ankylosis
  * Must have been previously exposed to 1 or 2 bDMARDs (at least 1 tumor necrosis factor [TNF] inhibitor or 1 interleukin [IL]-17 inhibitor [IL-17i]), and must have discontinued the bDMARD therapy due to either lack of efficacy (after at least 12 weeks of treatment with a bDMARD at an adequate dose) or intolerance (irrespective of treatment duration). Prior exposure to two bDMARDs was allowed for no more than 30% of patients; among patients with prior exposure to two bDMARDs, a lack of efficacy to one bDMARD and intolerance to another was permitted, but a patient could not have a lack of efficacy to two bDMARDs
* Study 2:

  * Must have a clinical diagnosis of nr-axSpA fulfilling the 2009 Assessment of SpondyloArthritis international Society (ASAS) classification criteria for axSpA but not meeting the radiologic criterion of the modified New York criteria for AS
  * Must have objective signs of active inflammation consistent with axSpA on magnetic resonance imaging (MRI) of sacroiliac (SI) joints or based on high sensitivity C-reactive protein (hsCRP) > the upper limit of normal (ULN).
  * Prior treatment with at most one bDMARD (either TNF inhibitor or IL-17i) is allowed for at least 20% but no more than 35% of enrolled patients who had to discontinue the prior bDMARD due to either lack of efficacy (after ≥ 12 weeks at an adequate dose) or intolerance (regardless of treatment duration).
* Must have a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4 at the Screening and Baseline Visits.
* Must have a Total Back Pain score ≥ 4 based on a 0 - 10 numerical rating scale at the Screening and Baseline Visits.
* Has had an inadequate response to at least 2 nonsteroidal anti-inflammatory drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or has an intolerance to or contraindication for NSAIDs as defined by the Investigator.

Exclusion Criteria:

* Must not have been exposed to any Janus kinase (JAK) inhibitor (including but not limited to upadacitinib [Rinvoq®], tofacitinib [Xeljanz®], baricitinib [Olumiant®], filgotinib, ruxolitinib [Jakafi®], abrocitinib [PF-04965842], and peficitinib [Smyraf®]).
* Prior bDMARD therapy must be washed out.
* Participant must not have a history of an allergic reaction or significant sensitivity to constituents of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2025-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (212):
- United States (41):
  - Arizona Arthritis & Rheumatology Associates, P.C. /ID# 215282, Flagstaff, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 215113, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 214731, Tucson, Arizona
  - Newport Huntington Medical Group /ID# 216281, Huntington Beach, California
  - Inland Rheum & Osteo Med Grp /ID# 215807, Upland, California
  - Denver Arthritis Clinic /ID# 215346, Denver, Colorado
  - Tekton Research /ID# 215054, Fort Collins, Colorado
  - Arthritis & Rheumatic Disease Specialties /ID# 215306, Aventura, Florida
  - Sweet Hope Research Specialty Inc /ID# 215931, Hialeah, Florida
  - Innovation Medical Research Center /ID# 216068, Palmetto Bay, Florida
  - Conquest Research /ID# 215804, Winter Park, Florida
  - Great Lakes Clinical Trials /ID# 215790, Chicago, Illinois
  - Greater Chicago Specialty Physicians /ID# 216213, Schaumburg, Illinois
  - Clinic of Robert Hozman/Clinical Investigation Specialists /ID# 215055, Skokie, Illinois
  - Klein and Associates MD /ID# 214767, Hagerstown, Maryland
  - Tufts Medical Center /ID# 215925, Boston, Massachusetts
  - Clinical Pharmacology Study Group /ID# 215293, Worcester, Massachusetts
  - Wayne State University Health Center /ID# 215930, Detroit, Michigan
  - Advanced Rheumatology, PC /ID# 214973, Lansing, Michigan
  - St. Paul Rheumatology /ID# 215537, Eagan, Minnesota
  - Clinvest Research LLC /ID# 215785, Springfield, Missouri
  - CenterPointe Institute of Research /ID# 215793, St Louis, Missouri
  - NYU Langone Orthopedic Center /ID# 215594, New York, New York
  - St. Lawrence Health System /ID# 215844, Potsdam, New York
  - Cape Fear Arthritis Care /ID# 215927, Leland, North Carolina
  - Marietta Memorial Hospital /ID# 215929, Marietta, Ohio
  - STAT Research, Inc. /ID# 215264, Springboro, Ohio
  - Health Research of Oklahoma /ID# 215117, Oklahoma City, Oklahoma
  - Oregon Health and Science University /ID# 216446, Portland, Oregon
  - Altoona Ctr Clinical Res /ID# 214770, Duncansville, Pennsylvania
  - Tekton Research, Inc. /ID# 214923, Austin, Texas
  - Trinity Universal Research Associates - Carrollton /ID# 214948, Carrollton, Texas
  - Arthritis and Osteoporosis Clinic Of Brazos Valley /ID# 215805, College Station, Texas
  - JPS Rheumatology Clinic /ID# 215962, Fort Worth, Texas
  - Memorial Rheumatology /ID# 216311, Houston, Texas
  - Biopharma Informatic, LLC /ID# 215885, Houston, Texas
  - Biopharma Informatic - Park Row /ID# 215907, Houston, Texas
  - West Texas Clinical Research /ID# 215928, Lubbock, Texas
  - Trinity Universal Research Associates, Inc /ID# 215189, Plano, Texas
  - Rheumatology and Pulmonary Clinic /ID# 214946, Beckley, West Virginia
  - West Virginia Research Inst /ID# 214921, South Charleston, West Virginia
- Argentina (7):
  - Organizacion Medica de Investigacion (OMI) /ID# 214557, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Centro de Enfermedades del Hígado y Aparato Digestivo /ID# 214556, Rosario, Santa Fe Province
  - Instituto CAICI /ID# 215242, Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas Tucuman /ID# 214559, San Miguel de Tucumán, Tucumán Province
  - Hospital Cordoba /ID# 215846, Córdoba
  - Instituto Medico Strusberg /ID# 215239, Córdoba
  - Cimer /Id# 215240, San Miguel de Tucumán
- Australia (5):
  - Emeritus Research Sydney /ID# 215507, Botany, New South Wales
  - BJC Health /ID# 215510, Paramatta, New South Wales
  - Emeritus Research /ID# 215506, Camberwell, Victoria
  - Monash Medical Centre /ID# 215509, Clayton, Victoria
  - Barwon Rheumatology Services /ID# 215508, Geelong, Victoria
- Belgium (3):
  - UZ Gent /ID# 215004, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 215006, Leuven, Vlaams-Brabant
  - ReumaClinic /ID# 215005, Genk
- Brazil (5):
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 215277, Juiz de Fora, Minas Gerais
  - EDUMED Educacao em Saude S/S L /ID# 215111, Curitiba, Paraná
  - LMK Sevicos Medicos S/S /ID# 215112, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto /ID# 215176, São José do Rio Preto, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas /ID# 215175, São Paulo
- Bulgaria (8):
  - UMHAT Kaspela EOOD /ID# 214803, Plovdiv
  - Medical center Unimed /ID# 214816, Plovdiv
  - MHAT Plovdiv /ID# 214815, Plovdiv
  - Medical center Teodora /ID# 214813, Rousse
  - Medical center Excelsior /ID# 214805, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 214804, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 214806, Sofia
  - Diagnostic consultative center 17 Sofia /ID# 214808, Sofia
- Canada (5):
  - Percuro Clinical Research, Ltd /ID# 215302, Victoria, British Columbia
  - Toronto Western Hospital /ID# 215041, Toronto, Ontario
  - Applied Medical Informatics Research Inc. (AMIR) /ID# 215303, Montreal, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 215096, Trois-Rivières, Quebec
  - Centre de recherche du CHUQ /ID# 215038, Québec
- China (11):
  - The first affiliated hospital of bengbu medical college /ID# 216609, Bengbu, Anhui
  - Anhui Provincial Hospital /ID# 216631, Hefei, Anhui
  - Peking Union Medical College Hospital /ID# 216545, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital /ID# 216645, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College /ID# 217883, Shantou, Guangdong
  - Shenzhen People's Hospital /ID# 225438, Shenzhen, Guangdong
  - Zhuzhou Central Hospital /ID# 216644, Zhuzhou, Hunan
  - The First Affiliated Hospital of BaoTou Medical College, Inner Mongolia Universi /ID# 216612, Baotou, Inner Mongolia
  - The First Affiliated Hospital of Soochow University /ID# 216607, Suzhou, Jiangsu
  - Huashan Hospital, Fudan University /ID# 216646, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University /ID# 217945, Kunming
- Czechia (11):
  - REVMACLINIC s.r.o. /ID# 215153, Brno
  - Revmacentrum MUDr. Mostera, s.r.o. /ID# 215161, Brno
  - Revmatologie, s.r.o. /ID# 215309, Brno
  - CCR Ostrava, s.r.o. /ID# 215226, Ostrava
  - ARTHROHELP, s.r.o. /ID# 215224, Pardubice
  - Revmatologicky ustav v Praze /ID# 215154, Prague
  - PV MEDICAL Services s.r.o. /ID# 215119, Prague
  - Revmatologicka ambulance - MUDr. Zuzana Urbanova /ID# 215652, Prague
  - Thomayerova nemocnice /ID# 215118, Prague
  - Fakultni Nemocnice v Motole /ID# 215160, Prague
  - MEDICAL PLUS, s.r.o. /ID# 215324, Uherské Hradiště
- France (4):
  - CHU Toulouse /ID# 214780, Toulouse, Occitanie
  - CHU Bordeaux - Hopital Pellegrin /ID# 214784, Bordeaux
  - Hopital Ambroise Pare /ID# 214783, Boulogne-Billancourt
  - AP-HP - Hopital Cochin /ID# 214782, Paris
- Germany (9):
  - Universitaetsklinikum Erlangen /ID# 214281, Erlangen, Bavaria
  - Rheumatologische Schwerpunktpraxis Brandt-Juergens /ID# 214282, Berlin
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 214211, Berlin
  - Rheuma Research Lausitz, Dr. Mario Sutowicz /ID# 214218, Cottbus
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 214207, Dresden
  - Praxisgemeinschaft Rheumatologie Nephrologie Erlangen /ID# 214212, Erlangen
  - MVZ Rheumatologie und Autoimmunmedizin Hamburg GmbH /ID# 214208, Hamburg
  - Medizinische Hochschule Hannover /ID# 214209, Hanover
  - MVZ für Rheumatologie Dr. M. Welcker GmbH /ID# 214261, Planegg
- Hungary (8):
  - Debreceni Egyetem Klinikai Kozpont /ID# 215187, Debrecen, Hajdú-Bihar
  - Vital Medical Center Orvosi es Fogaszati Kozpont /ID# 215182, Veszprém, Veszprém megye
  - Rehavita Kft HU /ID# 215188, Kormend, Zala County
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 215183, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz /ID# 215186, Gyula
  - Hevizgyogyfurdo es Szent Andras Reumakorhaz /ID# 215184, Hévíz
  - Pest Megyei Flor Ferenc Korhaz /ID# 214501, Kistarcsa
  - CMED Rehabilitacios es Diagnosztikai Kozpont /ID# 215181, Székesfehérvár
- Israel (4):
  - The Chaim Sheba Medical Center /ID# 215854, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 216956, Tel Aviv, Tel Aviv
  - Bnai Zion Medical Center /ID# 215856, Haifa
  - Meir Medical Center /ID# 217255, Kfar Saba
- Japan (16):
  - Daido Clinic /ID# 214735, Nagoya, Aichi-ken
  - Matsuyama Red Cross Hospital /ID# 216021, Matsuyama, Ehime
  - National Hospital Organization Asahikawa Medical Center /ID# 214930, Asahikawa-shi, Hokkaido
  - Hokkaido University Hospital /ID# 215221, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 214598, Kobe, Hyōgo
  - Hyogo College of Medicine College Hospital /Id# 215638, Nishinomiya-shi, Hyōgo
  - Kita-harima Medical Center /ID# 216069, Ono-shi, Hyōgo
  - Kuwana City Medical Center /ID# 215196, Kuwana-shi, Mie-ken
  - Nagasaki University Hospital /ID# 215947, Nagasaki, Nagasaki
  - Sasebo Chuo Hospital /ID# 214703, Sasebo-shi, Nagasaki
  - Japanese Red Cross Okayama Hospital /ID# 214732, Okayama, Okayama-ken
  - Okinawa Prefectural Chubu Hospital /ID# 215575, Uruma, Okinawa
  - National Hospital Organization Osaka Minami Medical Center /ID# 214205, Kawachinagano Shi, Osaka
  - Osaka City General Hospital /ID# 215640, Osaka, Osaka
  - Juntendo University Hospital /ID# 214929, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 215414, Chuo-ku, Tokyo
- CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 215217, Mexico City, Mexico City, Mexico
- New Zealand (2):
  - Middlemore Clinical Trials /ID# 215502, Papatoetoe, Auckland
  - Waikato Hospital /ID# 215503, Hamilton, Waikato Region
- Poland (6):
  - AI Centrum Medyczne Sp. z o.o. sp.k. /ID# 214354, Poznan, Greater Poland Voivodeship
  - Nasz Lekarz Przychodnie Medyczne /ID# 214352, Torun, Kuyavian-Pomeranian Voivodeship
  - WroMedica I. Bielicka, A. Strzalkowska s.c. /ID# 215093, Wroclaw, Lower Silesian Voivodeship
  - REUMED Sp.z o.o. Filia nr 1 /ID# 214353, Lublin, Lublin Voivodeship
  - Osteo-Medic S.C. /ID# 214351, Bialystok, Podlaskie Voivodeship
  - ETYKA-Osrodek Badan Klinicznych /ID# 215572, Olsztyn, Warmian-Masurian Voivodeship
- Russia (19):
  - Chelyabinsk Regional Clinical Hospital /ID# 214463, Chelyabinsk, Chelyabinsk Oblast
  - Immanuel Kant Baltic Federal University /ID# 218259, Kaliningrad, Kaliningrad Oblast
  - LLC Family Outpatient Clinic № /ID# 214455, Korolev, Moscow
  - Research Institute of Rheumatology named after V.A. Nasonova /ID# 214459, Moscow, Moscow
  - LLC Medical Center /ID# 214410, Novosibirsk, Novosibirsk Oblast
  - Nort-Western State Medical University n.a. Mechnikov /ID# 214454, Saint Petersburg, Sankt-Peterburg
  - LLC Novaya Klinika /ID# 214420, Pyatigorsk, Stavropol Kray
  - Family Clinic /ID# 214737, Yekaterinburg, Sverdlovsk Oblast
  - Central City Hospital #7 /ID# 214741, Yekaterinburg, Sverdlovsk Oblast
  - Kazan State Medical University /ID# 214421, Kazan', Tatarstan, Respublika
  - Alliance Biomedical Ural Group /ID# 214457, Izhevsk, Udmurtiya Republic
  - Olla-Med Clinic /ID# 214460, Moscow
  - City Clinical Hospital n.a. O.M. Filatov /ID# 214486, Moscow
  - Omsk Regional Clinic Hospital /ID# 214464, Omsk
  - Orenburg State Medical University /ID# 214408, Orenburg
  - Ryazan State Medical University named after academician I.P. Pavlov /ID# 214418, Ryazan
  - Clinical Rheumatologic Hospital No 25 /ID# 214488, Saint Petersburg
  - RZD-Medicine Saratov /ID# 214465, Saratov
  - Ulyanovsk Regional Clinical Hospital /ID# 214458, Ulyanovsk
- Slovakia (5):
  - Univerzitna nemocnica Bratislava Nemocnica Stare Mesto /ID# 214675, Bratislava
  - Reum.hapi s.r.o. /ID# 224268, Nové Mesto nad Váhom
  - Narodny ustav reumatickych chorob /ID# 214674, Piešťany
  - MUDr. Zuzana Cizmarikova s.r.o. /ID# 215220, Poprad
  - ALBAMED s.r.o. /ID# 215248, Zvolen
- South Korea (7):
  - Ajou University Hospital /ID# 214533, Suwon, Gyeonggido
  - Hanyang University Seoul Hospital /ID# 214297, Seoul, Seoul Teugbyeolsi
  - Gachon University Gil Medical Center /ID# 214534, Incheon
  - Seoul National University Hospital /ID# 214532, Seoul
  - Kyunghee University Hospital at Gangdong /ID# 214296, Seoul
  - Asan Medical Center /ID# 214294, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital /ID# 214295, Seoul
- Spain (7):
  - Hospital Marina Baixa /ID# 215970, Villajoyosa, Alicante
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 214967, Sabadell, Barcelona
  - Hospital Unversitario Marques de Valdecilla /ID# 214965, Santander, Cantabria
  - Hospital Meixoeiro (CHUVI) /ID# 214969, Vigo, Pontevedra
  - Hospital Universitario Reina Sofia /ID# 214968, Córdoba
  - Hospital Universitario La Paz /ID# 216032, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 214966, Valencia
- Taiwan (5):
  - Kaohsiung Veterans General Hos /ID# 214332, Kaohsiung City, Taichung
  - Far Eastern Memorial Hospital /ID# 215384, New Taipei City
  - Chung Shan Medical University Hospital /ID# 214018, Taichung
  - China Medical University Hospital /ID# 214019, Taichung
  - Cathay General Hospital /ID# 214183, Taipei
- Turkey (Türkiye) (3):
  - Hacettepe Universitesi Tip Fak /ID# 214898, Sihhiye, Ankara
  - Istanbul University Cerrahpasa Faculty of Medicine /ID# 214895, Cerrahpaşa
  - Mugla Sitki Kocman University Medical Faculty /ID# 215358, Muğla
- Ukraine (16):
  - MNPE Chernihiv Regional Hospital of the Chernihiv Region Council /ID# 214145, Chernihiv
  - State Institution L.T. Malaya Therapy National Institute of the NAMS of Ukraine /ID# 214155, Kharkiv
  - CNCE of Kharkiv Regional Council Regional Clinical Hospital /ID# 214158, Kharkiv
  - MNI City Multidisciplinary Hospital #18 /ID# 214154, Kharkiv
  - Khmelnytskyi Regional Hospital /ID# 214153, Khmelnytskyi
  - MI Kryvyi Rih City Clinical Hospital No.2 /ID# 214152, Kryvyi Rih
  - Medical Center LLC Institute of Rheumatology /ID# 214146, Kyiv
  - Kyiv Railway Clinical Hosp No.2 /ID# 214779, Kyiv
  - Medical Center CONSILIUM MEDICAL /ID# 216234, Kyiv
  - MNI KRC Kyiv Regional Clinical Hospital /ID# 214156, Kyiv
  - Municipal Non-Commercial Enterprise Odesa Regional Clinical Hospital of the Od /ID# 214159, Odesa
  - Multifield Medical Centre of ONMU /ID# 214149, Odesa
  - PI "Poltava Regional Clinical Hospital n.a. M.V.Sklifosovsky" /ID# 214151, Poltava
  - Ternopil University Hospital /ID# 214705, Ternopil
  - CNE Vinnytsya Regional Clinical Hospital named after N.I.Pirogov /ID# 214147, Vinnytsia
  - Clinic of Scientific Research Institute of Invalid Rehabilitation /ID# 214148, Vinnytsia
- United Kingdom (4):
  - Minerva Health Centre /ID# 216226, Preston, Lancashire
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 214865, Norwich, Norfolk
  - West Suffolk Hospital /ID# 215529, Bury St Edmunds, Suffolk
  - Doncaster Royal Infirmary /ID# 214971, Armthorpe Road

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Navarro-Compan V, Van den Bosch F, Sampaio-Barros PD, Ostor AJK, Parikh B, Kato K, Gao T, Stigler J, Ramiro S. Efficacy of upadacitinib in subgroups of patients with axial spondyloarthritis with early versus established disease. RMD Open. 2025 Mar 4;11(1):e005110. doi: 10.1136/rmdopen-2024-005110. PMID 40037923
- [Derived] Van den Bosch F, Deodhar A, Poddubnyy D, Maksymowych WP, van der Heijde D, Kim TH, Kishimoto M, Baraliakos X, Bu X, Lagunes-Galindo I, Song IH, Wung P, Kato K, Shmagel A. Upadacitinib in active non-radiographic axial spondyloarthritis: 2-year data from the phase 3 SELECT-AXIS 2 study. Arthritis Res Ther. 2025 Feb 4;27(1):23. doi: 10.1186/s13075-024-03441-3. PMID 39905436
- [Derived] Baraliakos X, van der Heijde D, Sieper J, Inman RD, Kameda H, Maksymowych WP, Lagunes-Galindo I, Bu X, Wung P, Kato K, Shmagel A, Deodhar A. Efficacy and safety of upadacitinib in patients with active ankylosing spondylitis refractory to biologic therapy: 2-year clinical and radiographic results from the open-label extension of the SELECT-AXIS 2 study. Arthritis Res Ther. 2024 Nov 12;26(1):197. doi: 10.1186/s13075-024-03412-8. PMID 39533349
- [Derived] Burmester GR, Stigler J, Rubbert-Roth A, Tanaka Y, Azevedo VF, Coombs D, Lagunes I, Lippe R, Wung P, Gensler LS. Safety Profile of Upadacitinib up to 5 Years in Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis: An Integrated Analysis of Clinical Trials. Rheumatol Ther. 2024 Jun;11(3):737-753. doi: 10.1007/s40744-024-00671-4. Epub 2024 Apr 29. PMID 38683479
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Kiltz U, Kishimoto M, Walsh JA, Sampaio-Barros P, Mittal M, Saffore CD, Wung P, Ganz F, Biljan A, Poddubnyy D. Effect of Upadacitinib on Quality of Life and Work Productivity in Active Non-radiographic Axial Spondyloarthritis: Results From Randomized Phase 3 Trial SELECT-AXIS 2. Rheumatol Ther. 2023 Aug;10(4):887-899. doi: 10.1007/s40744-023-00550-4. Epub 2023 May 16. PMID 37191738
- [Derived] Navarro-Compan V, Baraliakos X, Magrey M, Ostor A, Saffore CD, Mittal M, Song IH, Ganz F, Stigler J, Deodhar A. Effect of Upadacitinib on Disease Activity, Pain, Fatigue, Function, Health-Related Quality of Life and Work Productivity for Biologic Refractory Ankylosing Spondylitis. Rheumatol Ther. 2023 Jun;10(3):679-691. doi: 10.1007/s40744-023-00536-2. Epub 2023 Feb 23. PMID 36820984
- [Derived] Deodhar A, Van den Bosch F, Poddubnyy D, Maksymowych WP, van der Heijde D, Kim TH, Kishimoto M, Blanco R, Duan Y, Li Y, Pangan AL, Wung P, Song IH. Upadacitinib for the treatment of active non-radiographic axial spondyloarthritis (SELECT-AXIS 2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2022 Jul 30;400(10349):369-379. doi: 10.1016/S0140-6736(22)01212-0. PMID 35908570
- [Derived] van der Heijde D, Baraliakos X, Sieper J, Deodhar A, Inman RD, Kameda H, Zeng X, Sui Y, Bu X, Pangan AL, Wung P, Song IH. Efficacy and safety of upadacitinib for active ankylosing spondylitis refractory to biological therapy: a double-blind, randomised, placebo-controlled phase 3 trial. Ann Rheum Dis. 2022 Nov;81(11):1515-1523. doi: 10.1136/ard-2022-222608. Epub 2022 Jul 4. PMID 35788492
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This master protocol consists of 2 independent studies with a common screening platform for adults with active axial spondyloarthritis (axSpA). Study 1 enrolled adults with ankylosing spondylitis (AS) who had an inadequate response (IR) to biologic disease-modifying antirheumatic drug (bDMARD) therapy. Study 2 enrolled adults with non-radiographic axSpA (nr-axSpA).
  Each study includes a double-blind treatment period and an ongoing open-label extension period. Results are reported up to Week 52.
Pre-assignment Details: In each study participants were randomized equally to one of two treatment groups. In Study 1 randomization was stratified by high-sensitivity C-reactive protein (hsCRP) at Screening, class of the prior bDMARD use, and geographic region. In Study 2 randomization was stratified by magnetic resonance imaging (MRI) and Screening hsCRP status, and exposure to bDMARDs. For both studies Japan and China each had a separate randomization schedule stratified by Screening hsCRP and MRI (Study 2 only).
Groups:
- Study 1: Placebo / Upadacitinib 15 mg: Participants with bDMARD-inadequate response ankylosing spondylitis (bDMARD-IR AS) received placebo tablets orally once a day for 14 weeks. At Week 14 participants switched to receive 15 mg upadacitinib once a day in the open-label extension period.
- Study 1: Upadacitinib 15 mg / Upadacitinib 15 mg: Participants with bDMARD-IR AS received 15 mg upadacitinib orally once a day for 14 weeks. At Week 14 participants continued to receive 15 mg upadacitinib once a day in the open-label extension period.
- Study 2: Placebo: Participants with nr-axSpA received placebo orally once a day for 52 weeks.
- Study 2: Upadacitinib 15 mg: Participants with nr-axSpA received 15 mg upadacitinib orally once a day for 52 weeks.
Period: Week 1 to Week 14
Arm/Group | Study 1: Placebo / Upadacitinib 15 mg | Study 1: Upadacitinib 15 mg / Upadacitinib 15 mg | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Started (Randomized) | 209 | 211 | 158 | 156
Received Study Drug (Study drug refers to either upadacitinib or placebo) | 209 | 211 | 157 | 156
Completed (Completed Week 14) | 204 | 206 | 149 | 142
Not Completed | 5 | 5 | 9 | 14
Not completed — Adverse Event | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 5 | 6
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Coronavirus Disease of 2019 (COVID-19) Logistical Restrictions | 0 | 1 | 0 | 0
Not completed — Other | 1 | 3 | 3 | 5
Period: Week 14 to Week 52
Arm/Group | Study 1: Placebo / Upadacitinib 15 mg | Study 1: Upadacitinib 15 mg / Upadacitinib 15 mg | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Started | 204 | 206 | 149 | 142
Completed (Completed Week 52) | 192 | 194 (One participant who was ongoing at the Week 52 data cut off date (19 May 2022) completed their Week 52 visit shortly thereafter.) | 138 | 133
Not Completed | 12 | 12 | 11 | 9
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5 | 7 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1
Not completed — COVID-19 Logistical Restrictions | 1 | 0 | 0 | 0
Not completed — Other | 4 | 5 | 4 | 5
Not completed — Ongoing | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) includes all randomized participants who received at least one dose of study drug (upadacitinib or placebo).
Groups:
- Study 1: Placebo: Participants with bDMARD-IR AS received placebo tablets orally once a day for 14 weeks. At Week 14 participants switched to receive 15 mg upadacitinib once daily in the open-label extension period.
- Study 1: Upadacitinib 15 mg: Participants with bDMARD-IR AS received 15 mg upadacitinib orally once a day for 14 weeks and continued to receive 15 mg upadacitinib once daily from Week 14 in the open-label extension period.
- Study 2: Placebo: Participants with nr-axSpA received placebo tablets orally once a day for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg | Study 2: Placebo | Study 2: Upadacitinib 15 mg | Total
Number analyzed (Participants) | 209 | 211 | 157 | 156 | 733
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Results are reported separately for Study 1 and Study 2
  years
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1 | 42.2 (11.78) | 42.6 (12.39) |  |  | 42.4 (12.08)
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2 |  |  | 42.5 (12.44) | 41.6 (12.00) | 42.1 (12.21)
Age, Customized [Count of Participants; unit: Participants] — Population: Results are reported separately for Study 1 and Study 2
  Participants
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1: < 40 years | 92 | 87 |  |  | 179
    Study 1: 40 - < 65 years | 108 | 112 |  |  | 220
    Study 1: ≥ 65 years | 9 | 12 |  |  | 21
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2: < 40 years |  |  | 67 | 72 | 139
    Study 2: 40 - < 65 years |  |  | 84 | 81 | 165
    Study 2: ≥ 65 years |  |  | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Results are reported separately for Study 1 and Study 2
  Participants
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1: Female | 51 | 58 |  |  | 109
    Study 1: Male | 158 | 153 |  |  | 311
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2: Female |  |  | 94 | 89 | 183
    Study 2: Male |  |  | 63 | 67 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Results are reported separately for Study 1 and Study 2
  Participants
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1: Hispanic or Latino | 20 | 17 |  |  | 37
    Study 1: Not Hispanic or Latino | 189 | 194 |  |  | 383
    Study 1: Unknown or Not Reported | 0 | 0 |  |  | 0
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2: Hispanic or Latino |  |  | 15 | 24 | 39
    Study 2: Not Hispanic or Latino |  |  | 142 | 132 | 274
    Study 2: Unknown or Not Reported |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Results are reported separately for Study 1 and Study 2
  Participants
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Study 1: Asian | 37 | 42 |  |  | 79
    Study 1: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Study 1: Black or African American | 3 | 1 |  |  | 4
    Study 1: White | 169 | 168 |  |  | 337
    Study 1: More than one race | 0 | 0 |  |  | 0
    Study 1: Unknown or Not Reported | 0 | 0 |  |  | 0
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2: American Indian or Alaska Native |  |  | 0 | 1 | 1
    Study 2: Asian |  |  | 28 | 19 | 47
    Study 2: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Study 2: Black or African American |  |  | 1 | 2 | 3
    Study 2: White |  |  | 127 | 134 | 261
    Study 2: More than one race |  |  | 1 | 0 | 1
    Study 2: Unknown or Not Reported |  |  | 0 | 0 | 0
Region [Count of Participants; unit: Participants] — Asia includes China, Taiwan, South Korea, and Japan.
  Other includes Australia, Israel, and New Zealand. Population: Results are reported separately for Study 1 and Study 2
  Participants
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1: North America | 25 | 25 |  |  | 50
    Study 1: South/Central America | 14 | 13 |  |  | 27
    Study 1: Western Europe | 25 | 16 |  |  | 41
    Study 1: Eastern Europe | 98 | 109 |  |  | 207
    Study 1: Asia | 34 | 41 |  |  | 75
    Study 1: Other | 13 | 7 |  |  | 20
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2: North America |  |  | 19 | 26 | 45
    Study 2: South/Central America |  |  | 13 | 12 | 25
    Study 2: Western Europe |  |  | 19 | 24 | 43
    Study 2: Eastern Europe |  |  | 72 | 68 | 140
    Study 2: Asia |  |  | 27 | 19 | 46
    Study 2: Other |  |  | 7 | 7 | 14
Time Since AS / nr-axSpA Diagnosis [Mean (Standard Deviation); unit: years] — Population: Results are reported separately for Study 1 and Study 2
  years
    Study 1 - Duration since AS diagnosis: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1 - Duration since AS diagnosis | 7.5 (7.51) | 7.9 (7.54) |  |  | 7.7 (7.52)
    Study 2 - Duration since nr-axSpA diagnosis: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2 - Duration since nr-axSpA diagnosis |  |  | 4.4 (5.83) | 4.5 (5.54) | 4.4 (5.68)
Duration of AS / nr-axSpA Symptoms [Mean (Standard Deviation); unit: years] — Population: Participants with available data; Results are reported separately for Study 1 and Study 2.
  years
    Study 1 -Duration of AS symptoms: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1 -Duration of AS symptoms | 12.6 (9.29) | 12.9 (9.08) |  |  | 12.8 (9.18)
    Study 2 - Duration of nr-axSpA symptoms: number analyzed (Participants) | 0 | 0 | 156 | 155 | 311
    Study 2 - Duration of nr-axSpA symptoms |  |  | 9.2 (8.12) | 9.0 (7.86) | 9.1 (7.98)
Study 1: Class of Prior bDMARD Use [Count of Participants; unit: Participants] — Population: Class of prior bDMARD use was collected in Study 1 only.
  Participants
    number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    One tumor necrosis factor (TNF) inhibitor | 158 | 154 |  |  | 312
    One interleukin-17 (IL-17) inhibitor | 24 | 29 |  |  | 53
    Prior exposure to 2 bDMARDs | 26 | 28 |  |  | 54
    Missing (no prior bDMARD use) | 1 | 0 |  |  | 1
Study 2: Prior bDMARD Use [Count of Participants; unit: Participants] — Population: Prior exposure to bDMARDs (yes or no) was a stratification factor in Study 2 only.
  Participants
    number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Yes |  |  | 54 | 49 | 103
    No |  |  | 103 | 107 | 210
High-sensitivity C-reactive Protein (hsCRP) Level at Screening [Count of Participants; unit: Participants] — The Screening level of hsCRP was a randomization stratification factor. The hsCRP upper limit of normal (ULN) = 2.87 mg/L. Population: Results are reported separately for Study 1 and Study 2
  Participants
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1: > upper limit of normal | 163 | 165 |  |  | 328
    Study 1: ≤ upper limit of normal | 46 | 46 |  |  | 92
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2: > upper limit of normal |  |  | 126 | 123 | 249
    Study 2: ≤ upper limit of normal |  |  | 31 | 33 | 64
Spondyloarthritis Research Consortium of Canada (SPARCC) MRI Spine Score [Mean (Standard Deviation); unit: score on a scale] — For the SPARCC MRI assessment of the spine, 6 discovertebral units (DVU) representing the 6 most abnormal DVUs were selected to calculate the MRI Spine SPARCC score. For each of the 6 DVUs, 3 consecutive sagittal slices were assessed in 4 quadrants to evaluate the extent of inflammation in all 3 dimensions. Each quadrant was scored for the presence (1) or absence (0) of edema. If edema was present in at least one quadrant of a DVU slice, it was also scored for intensity and depth of the edema. The maximum (worst) overall score for all 6 DVUs is 108. Population: Participants with available data; Results are reported separately for Study 1 and Study 2.
  score on a scale
    Study 1: number analyzed (Participants) | 209 | 199 | 0 | 0 | 408
    Study 1 | 8.8 (12.52) | 10.7 (15.43) |  |  | 9.7 (14.05)
    Study 2: number analyzed (Participants) | 0 | 0 | 147 | 139 | 286
    Study 2 |  |  | 1.4 (3.72) | 2.7 (6.88) | 2.1 (5.52)
SPARCC MRI Sacroiliac Joint Score [Mean (Standard Deviation); unit: score on a scale] — In the SPARCC MRI assessment of the sacroiliac (SI) joints 6 consecutive sacroiliac joint image coronal slices representing the largest proportion of the synovial compartment of the SI joints were assessed for edema, intensity and depth of edema.
  Each SI joint (left and right) was divided into quadrants for a total of 8 SI scoring locations. Each quadrant was scored for the presence (1) or absence (0) of edema, intensity of edema, and depth.
  The total maximum (worst) score for all SI joints across 6 slices is 72. Population: Participants with available data; Results are reported separately for Study 1 and Study 2.
  score on a scale
    Study 1: number analyzed (Participants) | 202 | 199 | 0 | 0 | 401
    Study 1 | 5.6 (10.63) | 5.0 (10.80) |  |  | 5.3 (10.71)
    Study 2: number analyzed (Participants) | 0 | 0 | 148 | 142 | 290
    Study 2 |  |  | 3.5 (7.60) | 4.4 (8.74) | 3.9 (8.18)
Study 2: Magnetic Resonance Imaging (MRI) Inflammation Status [Count of Participants; unit: Participants] — MRI-positive is defined as active sacroiliitis according to the Assessment of SpondyloArthritis international Society/Outcome Measures in Rheumatology Clinical Trials (ASAS/OMERACT) definition. Population: MRI inflammation status was only collected in Study 2.
  Participants
    number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    MRI-positive |  |  | 66 | 70 | 136
    MRI-negative |  |  | 91 | 86 | 177
Study 2: MRI Inflammation and hsCRP Status [Count of Participants; unit: Participants] — MRI-positive is defined as active sacroiliitis according to the ASAS/OMERACT definition; The hsCRP upper limit of normal (ULN) = 2.87 mg/L. Randomization of treatment assignment in Study 2 was stratified by positivity for MRI inflammation in the sacroiliac joints and screening hsCRP status (MRI-positive and hsCRP-positive, MRI-positive and hsCRP-negative, and MRI-negative and hsCRP-positive). Population: MRI inflammation status was only collected in Study 2.
  Participants
    number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    MRI positive and hsCRP > ULN |  |  | 35 | 38 | 73
    MRI positive and hsCRP ≤ ULN |  |  | 31 | 32 | 63
    MRI negative and hsCRP > ULN |  |  | 91 | 86 | 177
Patient's Global Assessment of Disease Activity (PtGA) [Mean (Standard Deviation); unit: units on a scale] — Assessed by the participant using a numeric rating scale (NRS) ranging from 0 (No activity) to 10 (Severe activity). Population: Results are reported separately for Study 1 and Study 2.
  units on a scale
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1 | 7.2 (1.40) | 7.4 (1.48) |  |  | 7.3 (1.44)
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2 |  |  | 7.3 (1.38) | 7.0 (1.62) | 7.1 (1.51)
Patient's Assessment of Total Back Pain [Mean (Standard Deviation); unit: units on a scale] — Total back pain was assessed by the participant on a NRS from 0 (no pain) to 10 (most severe pain). Population: Results are reported separately for Study 1 and Study 2.
  units on a scale
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1 | 7.4 (1.43) | 7.5 (1.48) |  |  | 7.4 (1.46)
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2 |  |  | 7.3 (1.39) | 7.2 (1.55) | 7.3 (1.47)
Bath Ankylosing Spondylitis Functional Index [Mean (Standard Deviation); unit: score on a scale] — The Bath Ankylosing Spondylitis Functional Index (BASFI) is used to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities, each scored on a NRS ranging from 0 (easy to perform activity) to 10 (impossible to perform activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher scores indicating more functional limitations. Population: Results are reported separately for Study 1 and Study 2.
  score on a scale
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1 | 6.2 (1.87) | 6.3 (2.03) |  |  | 6.2 (1.95)
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2 |  |  | 6.0 (2.14) | 5.9 (2.08) | 5.9 (2.11)
Inflammation [Mean (Standard Deviation); unit: score on a scale] — Inflammation was measured by the mean of the two morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each assessed on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration). Population: Results are reported separately for Study 1 and Study 2.
  score on a scale
    Study 1: number analyzed (Participants) | 209 | 211 | 0 | 0 | 420
    Study 1 | 6.8 (1.55) | 6.9 (1.84) |  |  | 6.8 (1.70)
    Study 2: number analyzed (Participants) | 0 | 0 | 157 | 156 | 313
    Study 2 |  |  | 6.7 (1.67) | 6.6 (1.83) | 6.6 (1.75)

OUTCOME MEASURES:

1. Primary Outcome: Study 1: Percentage of Participants Achieving Assessment of SpondyloArthritis International Society 40 (ASAS40) Response at Week 14
Description: ASAS40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units) in the potential remaining domain:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Week 14
Population: Full analysis set; participants who discontinued study drug prior to Week 14 or with missing data for reasons other than COVID-19 were counted as non-responders (non-responder imputation); Missing data due to COVID-19 infection or logistical restriction was handled by multiple imputation (MI).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Study 1: Placebo: Participants with bDMARD-IR AS received placebo tablets orally once a day for 14 weeks.
- Study 1: Upadacitinib 15 mg: Participants with bDMARD-IR AS received 15 mg upadacitinib orally once a day for 14 weeks.
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
percentage of participants | 18.2 [13.0 to 23.4] | 44.5 [37.8 to 51.3]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Efficacy analyses and hypothesis testing including multiplicity adjustment were performed independently for Study 1 and Study 2; Test type: Superiority — To preserve the overall type I error rate at α = 0.05 level, a multiple testing procedure was used to test the primary and multiplicity-controlled secondary endpoints. Testing began with the primary endpoint using two-sided α = 0.05; significance could be claimed for a lower ranked endpoint only if the previous endpoints in the sequence met the requirement of significance; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) model adjusted by main stratification factor of screening hsCRP level (> ULN vs ≤ ULN); Response Rate Difference = 26.4, 95% CI 2-sided [17.9 to 34.9] — Response Rate Difference = Upadacitinib - Placebo

2. Primary Outcome: Study 2: Percentage of Participants Achieving an ASAS40 Response at Week 14
Description: as for outcome 1
Time Frame: Baseline and Week 14
Population: Full analysis set; participants who discontinued study drug prior to Week 14 or with missing data for reasons other than COVID-19 were counted as non-responders (non-responder imputation); Missing data due to COVID-19 infection or logistical restriction was handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Study 2: Placebo: Participants with nr-axSpA received placebo tablets orally once a day for 14 weeks.
- Study 2: Upadacitinib 15 mg: Participants with nr-axSpA received 15 mg upadacitinib orally once a day for 14 weeks.
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 22.5 [16.0 to 29.1] | 44.9 [37.1 to 52.7]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Efficacy analyses and hypothesis testing including multiplicity adjustment were performed independently for Study 1 and Study 2. Binary endpoints in Study 2 were analyzed using the Cochran-Mantel-Haenszel (CMH) test stratified by the main stratification factor of positivity for MRI inflammation in the sacroiliac joints and screening hsCRP status (MRI-positive and hsCRP > ULN vs MRI-positive and hsCRP ≤ ULN vs MRI-negative and hsCRP > ULN); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP status; Response Rate Difference = 22.2, 95% CI 2-sided [12.1 to 32.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; A post-hoc logistic regression adjusting for the main stratification factor of MRI and screening hsCRP status was conducted for the multiplicity-controlled binary endpoints assessed at Week 14; Test type: Other; Odds Ratio (OR) = 2.8, 95% CI 2-sided [1.7 to 4.5] — Upadacitinib : Placebo

3. Secondary Outcome: Study 1: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 14
Description: ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L.
  The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). A negative change from Baseline score indicates improvement in disease activity.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with at least one available change from Baseline value; a mixed-effect model repeat measurement (MMRM) analysis including all observed data up to Week 14 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
score on a scale | -0.49 [-0.62 to -0.37] | -1.52 [-1.64 to -1.39]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — To preserve the overall type I error rate at α=0.05 level, a multiple testing procedure was used to test the primary and multiplicity-controlled secondary endpoints. Testing began with the primary endpoint using two-sided α = 0.05; significance could be claimed for a lower ranked endpoint only if the previous endpoints in the sequence met the requirement of significance; p < 0.0001, Mixed-effect Model Repeated Measurement; MMRM model includes treatment, visit and treatment-by-visit interaction, screening hsCRP level (> ULN vs ≤ ULN) and Baseline value as covariate; Least Squares (LS) Mean Difference = -1.02, 95% CI 2-sided [-1.20 to -0.85] — Treatment difference = Upadacitinib - Placebo

4. Secondary Outcome: Study 1: Change From Baseline in Magnetic Resonance Imaging (MRI) Spondyloarthritis Research Consortium of Canada (SPARCC) Score for the Spine at Week 14
Description: In the SPARCC MRI assessment of the spine, the entire spine was evaluated for active inflammation (bone marrow edema). Six discovertebral units (DVU) representing the 6 most abnormal DVUs were selected to calculate the MRI Spine SPARCC score. For each of the 6 DVUs, 3 consecutive sagittal slices were assessed in 4 quadrants to evaluate the extent of inflammation in all three dimensions.
  Each quadrant was scored for the presence (1) or absence (0) of edema. If edema was present in at least one quadrant of a DVU slice, it was also scored for intensity and depth of the edema representing that slice: An additional score of 1 was assigned if an intense signal was seen in any quadrant on a DVU slice. Slices that included a lesion demonstrating continuous increased signal of depth ≥ 1 cm extending from the endplate were scored as an additional 1 per slice.
  The maximum (worst) overall score for all 6 DVUs is 108. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available change from Baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 186 | 181
score on a scale | -0.04 [-1.14 to 1.06] | -3.95 [-5.06 to -2.83]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, ANCOVA; ANCOVA model including treatment and screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -3.90, 95% CI 2-sided [-5.47 to -2.33] — Treatment difference = Upadacitinib - Placebo

5. Secondary Outcome: Study 1: Percentage of Participants With Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response at Week 14
Description: The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For Questions 1 to 5 (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
  A BASDAI 50 response is defined as improvement of 50% or more from Baseline in BASDAI score.
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
percentage of participants | 16.7 [11.7 to 21.8] | 43.1 [36.4 to 49.8]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) model adjusted by main stratification factor of screening hsCRP level (> ULN vs ≤ ULN); Response Rate Difference = 26.4, 95% CI 2-sided [18.0 to 34.8] — Response Rate Difference = Upadacitinib - Placebo

6. Secondary Outcome: Study 1: Percentage of Participants With an ASAS20 Response at Week 14
Description: ASAS20 response was defined as an improvement of ≥ 20% and an absolute improvement of ≥ 1 unit (on a scale of 0 to 10) from Baseline in at least 3 of the following 4 domains, with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 units [on a scale of 0 to 10]) in the remaining domain:
  * Patient's global assessment of disease activity, measured on a NRS from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the BASFI which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related BASDAI NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
percentage of participants | 38.3 [31.7 to 44.9] | 65.4 [59.0 to 71.8]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) model adjusted by main stratification factor of screening hsCRP level (> ULN vs ≤ ULN); Response Rate Difference = 27.1, 95% CI 2-sided [17.9 to 36.3] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Study 1: Percentage of Participants With ASDAS Inactive Disease at Week 14
Description: ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L.
  The overall score ranges from 0 with no defined upper score. ASDAS Inactive Disease is defined as an ASDAS score < 1.3.
Time Frame: Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
percentage of participants | 1.9 [0.1 to 3.8] | 12.8 [8.3 to 17.3]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) model adjusted by main stratification factor of screening hsCRP level (> ULN vs ≤ ULN); Response Rate Difference = 10.9, 95% CI 2-sided [6.0 to 15.8] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Study 1: Change From Baseline in Patient's Assessment of Total Back Pain at Week 14
Description: Participants assessed their total back pain during the last week on a 0 to 10 numerical rating scale (NRS), where 0 represents no pain and 10 represents most severe pain.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with at least one available change from Baseline value; a mixed-effect model repeat measurement analysis including all observed data up to Week 14 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
score on a scale | -1.47 [-1.77 to -1.16] | -3.00 [-3.30 to -2.70]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -1.53, 95% CI 2-sided [-1.96 to -1.11] — Treatment difference = Upadacitinib - Placebo

9. Secondary Outcome: Study 1: Change From Baseline in Patient's Assessment of Nocturnal Back Pain at Week 14
Description: Participants assessed the amount of back pain at night over the last week on a 0 to 10 NRS, where 0 represents no pain and 10 represents most severe pain.
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 208 | 211
score on a scale | -1.52 [-1.84 to -1.20] | -3.21 [-3.52 to -2.89]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -1.69, 95% CI 2-sided [-2.14 to -1.24] — Treatment difference = Upadacitinib - Placebo

10. Secondary Outcome: Study 1: Percentage of Participants With ASDAS Low Disease Activity at Week 14
Description: ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L.
  The overall score ranges from 0 with no defined upper score. ASDAS Low Disease Activity is defined as an ASDAS score < 2.1.
Time Frame: Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
percentage of participants | 10.1 [6.0 to 14.2] | 44.1 [37.4 to 50.8]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) model adjusted by main stratification factor of screening hsCRP level (> ULN vs ≤ ULN); Response Rate Difference = 34.0, 95% CI 2-sided [26.2 to 41.8] — Response Rate Difference = Upadacitinib - Placebo

11. Secondary Outcome: Study 1: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 14
Description: The Bath Ankylosing Spondylitis Functional Index is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities such as putting on socks, bending, reaching, getting up from the floor or an armless chair, standing, climbing and other physical activities. Each item is scored on a NRS ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher scores indicating more functional limitations. A negative change from Baseline in BASFI indicates improvement.
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
score on a scale | -1.09 [-1.35 to -0.83] | -2.26 [-2.53 to -2.00]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -1.17, 95% CI 2-sided [-1.55 to -0.80] — Treatment difference = Upadacitinib - Placebo

12. Secondary Outcome: Study 1: Percentage of Participants With ASAS Partial Remission at Week 14
Description: ASAS partial remission (PR) is defined as an absolute score of ≤ 2 units on a 0 to 10 scale for each of the four following domains:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 209 | 211
percentage of participants | 4.3 [1.6 to 7.1] | 17.5 [12.4 to 22.7]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) model adjusted by main stratification factor of screening hsCRP level (> ULN vs ≤ ULN); Response Rate Difference = 13.2, 95% CI 2-sided [7.4 to 19.0] — Response Rate Difference = Upadacitinib - Placebo

13. Secondary Outcome: Study 1: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score at Week 14
Description: The ASQoL consists of 18 items related to quality of life, including the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. Each item is answered as yes (scored as 1) or no (scored as 0).
  Scores are summed to obtain the overall score which ranges from 0 to 18, where higher scores indicate a worse quality of life. A negative change from Baseline in ASQoL indicates improvement in quality of life.
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 208 | 210
score on a scale | -2.03 [-2.62 to -1.44] | -5.10 [-5.69 to -4.52]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -3.07, 95% CI 2-sided [-3.90 to -2.24] — Treatment difference = Upadacitinib - Placebo

14. Secondary Outcome: Study 1: Change From Baseline in ASAS Health Index at Week 14
Description: The ASAS health index (HI) measures functioning and health across 17 aspects of health in patients with AS, including pain, emotional functions, sleep, sexual function, mobility, self care, and community life. Each of the 17 questions is answered by the participant as "I agree" (score = 1) or "I disagree" (score = 0). The responses to the 17 dichotomous items are summed up to give a total score ranging from 0 to 17, where a higher score indicates a worse health status. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 208 | 211
score on a scale | -1.07 [-1.51 to -0.64] | -2.93 [-3.36 to -2.50]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -1.85, 95% CI 2-sided [-2.47 to -1.24] — Treatment difference = Upadacitinib - Placebo

15. Secondary Outcome: Study 1: Change From Baseline in Linear Bath Ankylosing Spondylitis Metrology Index (BASMI[Lin]) at Week 14
Description: The BASMI is a composite score based on 5 direct measurements of spinal mobility:
  1. cervical rotation (measured in degrees),
  2. tragus to wall distance (in centimeters [cm])
  3. lumbar side flexion (in cm),
  4. lumbar flexion (modified Schober's) (in cm) and
  5. intermalleolar distance (in cm).
  Each measurement is converted to a linear score between 0 and 10. The total BASMI(lin) score is the average of the 5 scores and ranges from 0 to 10; the higher the BASMI(lin) score the more severe the patient's limitation of movement due to their ankylosing spondylitis. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available change from Baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 201 | 205
score on a scale | -0.16 [-0.26 to -0.06] | -0.48 [-0.58 to -0.38]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, ANCOVA; ANCOVA model including treatment and screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -0.32, 95% CI 2-sided [-0.46 to -0.18] — Treatment difference = Upadacitinib - Placebo

16. Secondary Outcome: Study 1: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 14
Description: The MASES evaluation was conducted to assess the presence or absence of enthesitis (inflammation of the entheses, or sites where tendons or ligaments insert into the bone) at 13 different sites (first costochondral joint left/right, seventh costochondral joint left/right, posterior superior iliac spine left/right, anterior superior iliac spine left/right, iliac crest left/right, fifth lumbar spinous process, and proximal insertion of Achilles tendon left/right. Each site was scored for presence (1) or absence (0) of enthesitis. The MASES is the sum of the 13 site scores, and ranges from 0 to 13, with higher scores indicating more inflammation of the entheses. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with Baseline enthesitis and at least one available change from Baseline value; a mixed-effect model repeat measurement analysis including all observed data up to Week 14 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 162 | 148
score on a scale | -1.1 [-1.5 to -0.8] | -2.6 [-3.0 to -2.2]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.0 to -0.9] — Treatment difference = Upadacitinib - Placebo

17. Secondary Outcome: Study 1: Change From Baseline in MRI SPARCC Score for Sacroiliac Joints at Week 14
Description: In the SPARCC MRI assessment of the sacroiliac (SI) joints 6 consecutive sacroiliac joint image coronal slices representing the largest proportion of the synovial compartment of the SI joints were assessed for edema, intensity and depth of edema.
  Each SI joint (left and right) was divided into quadrants for a total of 8 SI scoring locations. Each quadrant was scored for the presence (1) or absence (0) of edema, intensity of edema (a score of 1 was assigned for each SI joint (left and right) if an intense signal was seen in any quadrant of that joint for each slice), and a lesion was graded as deep (score of 1) if there was homogeneous and unequivocal increase in signal extending over a depth of at least 1 cm from the articular surface of the SI joint in any quadrant.
  The total maximum (worst) score for all SI joints across 6 slices is 72. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available change from Baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: Upadacitinib 15 mg
Number analyzed (Participants) | 186 | 181
score on a scale | 1.05 [0.22 to 1.89] | -2.26 [-3.10 to -1.41]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: Upadacitinib 15 mg; Test type: Other; p < 0.0001, ANCOVA — This comparison was not part of the pre-specified multiplicity testing sequence; ANCOVA model including treatment and screening hsCRP level as fixed factors and Baseline value as covariate; LS Mean Difference = -3.31, 95% CI 2-sided [-4.50 to -2.12] — Treatment difference = Upadacitinib - Placebo

18. Secondary Outcome: Study 2: Change From Baseline in ASDAS at Week 14
Description: as for outcome 3
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 156 | 154
score on a scale | -0.71 [-0.85 to -0.56] | -1.36 [-1.50 to -1.21]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; MMRM model includes treatment, visit, treatment-by-visit interaction, main stratification factors MRI and screening hsCRP status, and Baseline value; LS Mean Difference = -0.65, 95% CI 2-sided [-0.85 to -0.45] — Treatment difference = Upadacitinib - Placebo

19. Secondary Outcome: Study 2: Change From Baseline in MRI SPARCC Score for SI Joints at Week 14
Description: as for outcome 17
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available change from Baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 148 | 140
score on a scale | 0.57 [-0.17 to 1.30] | -2.49 [-3.22 to -1.77]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, ANCOVA; ANCOVA model including treatment, main stratification factor, treatment and stratification factor interaction and Baseline value as covariate; LS Mean Difference = -3.06, 95% CI 2-sided [-4.08 to -2.04] — Treatment difference = Upadacitinib - Placebo

20. Secondary Outcome: Study 2: Percentage of Participants With BASDAI 50 Response at Week 14
Description: as for outcome 5
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 22.1 [15.5 to 28.6] | 42.3 [34.6 to 50.1]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 20.1, 95% CI 2-sided [10.1 to 30.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; [analysis description as in outcome 2, analysis 2]; Test type: Other; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.6 to 4.2] — Upadacitinib : Placebo

21. Secondary Outcome: Study 2: Percentage of Participants With ASDAS Inactive Disease at Week 14
Description: as for outcome 7
Time Frame: Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 5.2 [1.7 to 8.7] | 14.1 [8.6 to 19.6]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0063, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 8.8, 95% CI 2-sided [2.5 to 15.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; [analysis description as in outcome 2, analysis 2]; Test type: Other; Odds Ratio (OR) = 3.0, 95% CI 2-sided [1.3 to 7.0] — Upadacitinib : Placebo

22. Secondary Outcome: Study 2: Change From Baseline in Patient's Assessment of Total Back Pain at Week 14
Description: as for outcome 8
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 156 | 154
score on a scale | -2.00 [-2.35 to -1.65] | -2.91 [-3.27 to -2.56]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0004, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 18, analysis 1]; LS Mean Difference = -0.92, 95% CI 2-sided [-1.42 to -0.41] — Treatment difference = Upadacitinib - Placebo

23. Secondary Outcome: Study 2: Change From Baseline in Patient's Assessment of Nocturnal Back Pain at Week 14
Description: as for outcome 9
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 154 | 151
score on a scale | -1.84 [-2.23 to -1.44] | -2.96 [-3.36 to -2.56]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 18, analysis 1]; LS Mean Difference = -1.12, 95% CI 2-sided [-1.68 to -0.55] — Treatment difference = Upadacitinib - Placebo

24. Secondary Outcome: Study 2: Percentage of Participants With ASDAS Low Disease Activity at Week 14
Description: as for outcome 10
Time Frame: Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 18.3 [12.2 to 24.4] | 42.3 [34.6 to 50.1]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 23.8, 95% CI 2-sided [14.2 to 33.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; [analysis description as in outcome 2, analysis 2]; Test type: Other; Odds Ratio (OR) = 3.2, 95% CI 2-sided [1.9 to 5.4] — Upadacitinib : Placebo

25. Secondary Outcome: Study 2: Percentage of Participants With ASAS Partial Remission at Week 14
Description: as for outcome 12
Time Frame: Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 7.6 [3.5 to 11.8] | 18.6 [12.5 to 24.7]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0035, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 10.9, 95% CI 2-sided [3.6 to 18.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; [analysis description as in outcome 2, analysis 2]; Test type: Other; Odds Ratio (OR) = 2.7, 95% CI 2-sided [1.3 to 5.6] — Upadacitinib : Placebo

26. Secondary Outcome: Study 2: Change From Baseline in BASFI at Week 14
Description: as for outcome 11
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 156 | 154
score on a scale | -1.47 [-1.79 to -1.15] | -2.61 [-2.94 to -2.29]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 18, analysis 1]; LS Mean Difference = -1.14, 95% CI 2-sided [-1.60 to -0.68] — Treatment difference = Upadacitinib - Placebo

27. Secondary Outcome: Study 2: Change From Baseline in ASQoL at Week 14
Description: as for outcome 13
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 154 | 151
score on a scale | -3.15 [-3.87 to -2.43] | -5.38 [-6.11 to -4.65]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 18, analysis 1]; LS Mean Difference = -2.23, 95% CI 2-sided [-3.26 to -1.21] — Treatment difference = Upadacitinib - Placebo

28. Secondary Outcome: Study 2: Change From Baseline in ASAS Health Index at Week 14
Description: The ASAS HI measures functioning and health across 17 aspects of health in patients with AS, including pain, emotional functions, sleep, sexual function, mobility, self care, and community life. Each of the 17 questions is answered by the participant as "I agree" (score = 1) or "I disagree" (score = 0). The responses to the 17 dichotomous items are summed up to give a total score ranging from 0 to 17, where a higher score indicates a worse health status. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 154 | 150
score on a scale | -1.48 [-2.02 to -0.93] | -3.26 [-3.81 to -2.70]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 18, analysis 1]; LS Mean Difference = -1.78, 95% CI 2-sided [-2.56 to -1.00] — Treatment difference = Upadacitinib - Placebo

29. Secondary Outcome: Study 2: Percentage of Participants Achieving an ASAS20 Response at Week 14
Description: as for outcome 6
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 43.8 [36.0 to 51.5] | 66.7 [59.3 to 74.1]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 22.8, 95% CI 2-sided [12.2 to 33.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; [analysis description as in outcome 2, analysis 2]; Test type: Other; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.6 to 4.0] — Upadacitinib : Placebo

30. Secondary Outcome: Study 2: Change From Baseline in BASMI(Lin) at Week 14
Description: as for outcome 15
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available change from Baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 148 | 144
score on a scale | -0.19 [-0.29 to -0.08] | -0.29 [-0.40 to -0.18]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1781, ANCOVA; ANCOVA model including treatment and main stratification factor MRI and hsCRP status as fixed factors and Baseline value as covariate; LS Mean Difference = -0.10, 95% CI 2-sided [-0.25 to 0.05] — Treatment difference = Upadacitinib - Placebo

31. Secondary Outcome: Study 2: Change From Baseline in MASES at Week 14
Description: as for outcome 16
Time Frame: Baseline and Week 14
Population: as for outcome 16
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 125 | 124
score on a scale | -1.6 [-2.0 to -1.2] | -2.3 [-2.7 to -1.9]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Other; p = 0.0193, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 18, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.3 to -0.1] — Treatment difference = Upadacitinib - Placebo

32. Secondary Outcome: Study 2: Percentage of Participants Achieving an ASAS40 Response at Week 52
Description: as for outcome 1
Time Frame: Baseline and Week 52
Population: Full analysis set; participants who discontinued study drug prior to Week 52 or with missing data for reasons other than COVID-19 were counted as non-responders (non-responder imputation); Missing data due to COVID-19 infection or logistical restriction was handled by multiple imputation.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 42.7 [34.9 to 50.4] | 62.8 [55.2 to 70.4]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 20.1, 95% CI 2-sided [9.3 to 30.9] — Response Rate Difference = Upadacitinib - Placebo

33. Secondary Outcome: Study 2: Change From Baseline in MRI SPARCC Score for the Spine at Week 14
Description: In the SPARCC MRI assessment of the spine, the entire spine is evaluated for active inflammation (bone marrow edema). Six discovertebral units (DVU) representing the 6 most abnormal DVUs were selected to calculate the MRI Spine SPARCC score. For each of the 6 DVUs, 3 consecutive sagittal slices were assessed in 4 quadrants to evaluate the extent of inflammation in all three dimensions.
  Each quadrant was scored for the presence (1) or absence (0) of edema. If edema was present in at least one quadrant of a DVU slice, it was also scored for intensity and depth of the edema representing that slice: An additional score of 1 was assigned if an intense signal was seen in any quadrant on a DVU slice. Slices that included a lesion demonstrating continuous increased signal of depth ≥ 1 cm extending from the endplate were scored as an additional 1 per slice.
  The maximum (worst) overall score for all 6 DVUs is 108. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 14
Population: Full analysis set participants with available change from Baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 146 | 136
score on a scale | 0.34 [-0.32 to 1.00] | -0.79 [-1.48 to -0.11]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Other; p = 0.0206, ANCOVA — This comparison was not part of the pre-specified multiplicity testing sequence; ANCOVA model including treatment and main stratification factors MRI and hsCRP status as fixed factors and Baseline value as covariate; LS Mean Difference = -1.13, 95% CI 2-sided [-2.08 to -0.17] — Treatment difference = Upadacitinib - Placebo

34. Secondary Outcome: Study 2: Percentage of Participants Who Initiated Rescue Treatment Between Week 24 and Week 52
Description: Participants who did not achieve an ASAS20 response at any 2 consecutive scheduled visits from Week 24 through Week 52 were to be rescued with standard of care treatment as described in the protocol.
Time Frame: Week 24, Week 32, Week 40, and Week 52
Population: The analysis population is the Full Analysis Set, which includes all participants who were randomized and received at least one dose of study drug. Even though rescue was not assessed until after Week 24, the interpretation of the analysis is based on the percentage of participants who were rescued out of those who were randomized and received study drug, similar to the analysis of other binary endpoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants
  Week 24 | 13.4 [8.5 to 19.7] | 5.1 [2.2 to 9.9]
  Week 32 | 1.9 [0.4 to 5.5] | 3.2 [1.0 to 7.3]
  Week 40 | 0.6 [0.0 to 3.5] | 0.6 [0.0 to 3.5]
  Week 52 | 1.3 [0.2 to 4.5] | 0 [0.0 to 2.3]

35. Secondary Outcome: Study 2: Percentage of Participants With ASDAS Major Improvement at Week 52
Description: ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L.
  The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). Major Improvement is defined as a change from Baseline of ≤ -2.0.
Time Frame: Baseline and Week 52
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 20.4 [14.1 to 26.7] | 37.8 [30.2 to 45.4]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 17.6, 95% CI 2-sided [7.9 to 27.3] — Response Rate Difference = Upadacitinib - Placebo

36. Secondary Outcome: Study 2: Percentage of Participants With ASDAS Inactive Disease at Week 52
Description: as for outcome 7
Time Frame: Week 52
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 10.8 [6.0 to 15.7] | 32.7 [25.3 to 40.1]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 21.9, 95% CI 2-sided [13.2 to 30.6] — Response Rate Difference = Upadacitinib - Placebo

37. Secondary Outcome: Study 2: Percentage of Participants With ASDAS Low Disease Activity at Week 52
Description: as for outcome 10
Time Frame: Week 52
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study 2: Placebo | Study 2: Upadacitinib 15 mg
Number analyzed (Participants) | 157 | 156
percentage of participants | 32.5 [25.2 to 39.9] | 55.8 [48.0 to 63.6]
Statistical Analysis 1: Comparison: Study 2: Placebo vs Study 2: Upadacitinib 15 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test stratified by main stratification factor of MRI and screening hsCRP level status; Response Rate Difference = 23.1, 95% CI 2-sided [12.4 to 33.7] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 14 (Study 1 Week 1 - 14 groups) or Week 52 (for Study 1 Week 1 - 52 and Study 2 groups)
Groups:
- Study 1 Week 1 - 14: Placebo: Participants with bDMARD-IR AS received placebo tablets orally once a day for 14 weeks.
- Study 1 Week 1 - 14: Upadacitinib 15 mg: Participants with bDMARD-IR AS received 15 mg upadacitinib orally once a day for 14 weeks.
- Study 1 Week 1 - 52: Upadacitinib 15 mg: Participants with bDMARD-IR AS originally assigned to placebo received 15 mg upadacitinib from Week 14 to Week 52 and participants originally assigned to upadacitinib received 15 mg upadacitinib from Week 1 to Week 52.
- Study 2 Week 1 - 52: Placebo: Participants with nr-axSpA received placebo tablets orally once a day for 52 weeks.
- Study 2 Week 1 - 52: Upadacitinib 15 mg: Participants with nr-axSpA received 15 mg upadacitinib orally once a day for 52 weeks.
Arm/Group | Study 1 Week 1 - 14: Placebo | Study 1 Week 1 - 14: Upadacitinib 15 mg | Study 1 Week 1 - 52: Upadacitinib 15 mg | Study 2 Week 1 - 52: Placebo | Study 2 Week 1 - 52: Upadacitinib 15 mg
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/211 | 1/414 | 0/157 | 0/156
Serious Adverse Events (participants affected / at risk) | 1/209 | 6/211 | 43/414 | 6/157 | 6/156
Other Adverse Events (participants affected / at risk) | 15/209 | 19/211 | 96/414 | 40/157 | 36/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 1 Week 1 - 14: Placebo (N=209) | Study 1 Week 1 - 14: Upadacitinib 15 mg (N=211) | Study 1 Week 1 - 52: Upadacitinib 15 mg (N=414) | Study 2 Week 1 - 52: Placebo (N=157) | Study 2 Week 1 - 52: Upadacitinib 15 mg (N=156)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IRIDOCYCLITIS (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OPHTHALMOPLEGIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
REFRACTION DISORDER (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STRABISMUS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UVEITIS (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATIC CYST (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 4 (4) | 10 (10) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COMPLICATED APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DISSEMINATED VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGIC FEVER WITH RENAL SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TONSIL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 1 Week 1 - 14: Placebo (N=209) | Study 1 Week 1 - 14: Upadacitinib 15 mg (N=211) | Study 1 Week 1 - 52: Upadacitinib 15 mg (N=414) | Study 2 Week 1 - 52: Placebo (N=157) | Study 2 Week 1 - 52: Upadacitinib 15 mg (N=156)
COVID-19 (Infections and infestations) | 5 (5) | 6 (6) | 47 (48) | 21 (21) | 19 (19)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 5 (5) | 23 (35) | 8 (8) | 12 (15)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 2 (3) | 22 (30) | 8 (9) | 7 (8)
HEADACHE (Nervous system disorders) | 3 (3) | 7 (7) | 15 (16) | 6 (6) | 10 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT04169373/Prot_003.pdf
  • Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT04169373/SAP_001.pdf